CLINICAL TRIAL: NCT05858554
Title: The Safety of Direct Laparoscopic Introduction: Retrospective Observational Study at the University Hospital of Strasbourg
Acronym: Coelios
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8952
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-05

CONDITIONS: Laparoscopy
Keywords: Laparoscopy; coelioscopie; Veress Needle Technique

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Veress techniques and open laparoscopy are the techniques most used by gynecological surgeons to date. Advantages of the direct introduction unknown because technique still little used.

The research hypothesis is that very few major complications are expected showing the safety of direct introduction.

A look back at the practice of direct introduction into laparoscopy from 2012 to 2022 at the CMCO (Medical-Surgical and Obstetrical Center of Strasbourg)

ELIGIBILITY:
Inclusion criteria:

* Adult woman who had a scheduled or emergency laparoscopy at the CMCO between 01/01/2010 and 12/31/2022.
* Subject, having not expressed their opposition to the reuse of data of their data for the purposes of scientific research.

Exclusion criteria:

- Subject having expressed its opposition to the reuse of its data for scientific res

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman who had a scheduled or emergency laparoscopy at the CMCO between 01/01/2010 and 12/31/2022.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-12-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Study of intraoperative complications of direct introduction in open laparoscopy | Files analysed retrospectively from from January 01, 2010 to December 31, 2022 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie Obstétrique - CHU de Strasbourg - France, Strasbourg, France